CLINICAL TRIAL: NCT01846442
Title: Topical DHEA Against Vaginal Atrophy (3-Month Placebo-Controlled Double-Blind Randomized Phase III Study)
Brief Title: Topical DHEA Against Vaginal Atrophy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: EndoCeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ERC-210
Record Dates: First submitted 2013-05-01; First posted 2013-05-03 (Estimated); Results first posted 2017-04-28 (Actual); Last update posted 2017-08-29 (Actual); Status verified 2017-07

CONDITIONS: Vaginal Atrophy
Keywords: Vulvar/vaginal atrophy; Atrophic Vaginitis; Dehydroepiandrosterone; DHEA; Prasterone; Vaginorm; Menopause; Intrarosa
MeSH Terms: conditions — Atrophic Vaginitis | interventions — Dehydroepiandrosterone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- 0.25% DHEA (Experimental)
  Interventions: Drug: DHEA (0.25%)
- 0.5% DHEA (Experimental)
  Interventions: Drug: DHEA (0.5%)
- 1.0% DHEA (Experimental)
  Interventions: Drug: DHEA (1.0%)

INTERVENTIONS:
Drug: Placebo — Placebo vaginal suppository containing 0.0% (0 mg) DHEA; daily dosing with one suppository for 12 weeks.
  Other Names: Prasterone, Dehydroepiandrosterone
  Arms: Placebo
Drug: DHEA (0.25%) — Vaginal suppository containing 0.25% (3.25 mg) DHEA; daily dosing with one suppository for 12 weeks.
  Other Names: Prasterone, Dehydroepiandrosterone
  Arms: 0.25% DHEA
Drug: DHEA (0.5%) — Vaginal suppository containing 0.5% (6.5 mg) DHEA; daily dosing with one suppository for 12 weeks.
  Other Names: Prasterone, Dehydroepiandrosterone
  Arms: 0.5% DHEA
Drug: DHEA (1.0%) — Vaginal suppository containing 1.0% (13 mg) DHEA; daily dosing with one suppository for 12 weeks.
  Other Names: Prasterone, Dehydroepiandrosterone
  Arms: 1.0% DHEA

SUMMARY:
The purpose of this study is to determine the dose-response of vaginal mucosa parameters to the local action of DHEA (Dehydroepiandrosterone) in postmenopausal women suffering from vaginal atrophy.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women (non hysterectomized or hysterectomized)
* Women between 40 and 75 years of age
* Willing to participate in the study and sign an informed consent
* Women having a low maturation index (no greater part of guidance than 5% of superficial cells on vaginal smear)
* Women having a vaginal pH above 5
* Women who have self-identified at least one moderate to severe symptoms of vulvovaginal atrophy

Exclusion Criteria:

* Undiagnosed abnormal genital bleeding
* Hypertension equal to or above 160/95 mm Hg or not controlled by standard therapy
* The administration of any investigational drug within 30 days of screening visit
* Endometrial hyperplasia at biopsy performed at screening or endometrial cancer
* Use of estrogens/progestins products (vaginal, oral, pellet, transdermal, etc) in the 4 weeks to 6 months (depending on the product used) prior study entry

Ages: 40 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Actual)
Dates: Start 2007-06; Primary Completion 2008-05 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David F Archer, MD, Principal Investigator — Clinical Research Center, Eastern Virginia Medical Scholl, Norfolk, VA
Locations (8):
- United States (2):
  - EndoCeutics site # 05, Cleveland, Ohio
  - EndoCeutics site # 03, Norfolk, Virginia
- Canada (6):
  - EndoCeutics site # 10, Montreal, Quebec
  - EndoCeutics site # 09, Montreal, Quebec
  - EndoCeutics site # 08, Shawinigan, Quebec
  - EndoCeutics site # 11, Sherbrooke, Quebec
  - EndoCeutics site # 02, Québec
  - EndoCeutics site # 01, Québec

REFERENCES:
- [Result] Labrie F, Archer D, Bouchard C, Fortier M, Cusan L, Gomez JL, Girard G, Baron M, Ayotte N, Moreau M, Dube R, Cote I, Labrie C, Lavoie L, Berube R, Belanger P, Berger L, Gilbert L, Martel C, Balser J. Serum steroid levels during 12-week intravaginal dehydroepiandrosterone administration. Menopause. 2009 Sep-Oct;16(5):897-906. doi: 10.1097/gme.0b013e31819e8930. PMID 19436226
- [Result] Labrie F, Archer D, Bouchard C, Fortier M, Cusan L, Gomez JL, Girard G, Baron M, Ayotte N, Moreau M, Dube R, Cote I, Labrie C, Lavoie L, Berger L, Gilbert L, Martel C, Balser J. Intravaginal dehydroepiandrosterone (Prasterone), a physiological and highly efficient treatment of vaginal atrophy. Menopause. 2009 Sep-Oct;16(5):907-22. doi: 10.1097/gme.0b013e31819e8e2d. PMID 19436225
- [Result] Labrie F, Archer D, Bouchard C, Fortier M, Cusan L, Gomez JL, Girard G, Baron M, Ayotte N, Moreau M, Dube R, Cote I, Labrie C, Lavoie L, Berger L, Gilbert L, Martel C, Balser J. Effect of intravaginal dehydroepiandrosterone (Prasterone) on libido and sexual dysfunction in postmenopausal women. Menopause. 2009 Sep-Oct;16(5):923-31. doi: 10.1097/gme.0b013e31819e85c6. PMID 19424093
- [Result] Labrie F, Archer D, Bouchard C, Fortier M, Cusan L, Gomez JL, Girard G, Baron M, Ayotte N, Moreau M, Dube R, Cote I, Labrie C, Lavoie L, Berger L, Martel C, Balser J. High internal consistency and efficacy of intravaginal DHEA for vaginal atrophy. Gynecol Endocrinol. 2010 Jul;26(7):524-32. doi: 10.3109/09513590903511547. PMID 20459349
- [Result] Labrie F, Archer DF, Bouchard C, Fortier M, Cusan L, Gomez JL, Girard G, Baron M, Ayotte N, Moreau M, Dube R, Cote I, Labrie C, Lavoie L, Berger L, Gilbert L, Martel C, Balser J. Intravaginal dehydroepiandrosterone (prasterone), a highly efficient treatment of dyspareunia. Climacteric. 2011 Apr;14(2):282-8. doi: 10.3109/13697137.2010.535226. Epub 2011 Jan 18. PMID 21244215
- [Result] Labrie F, Archer D, Bouchard C, Fortier M, Cusan L, Gomez JL, Girard G, Baron M, Ayotte N, Moreau M, Dube R, Cote I, Labrie C, Lavoie L, Gilbert L, Martel C, Balser J. Lack of influence of dyspareunia on the beneficial effect of intravaginal prasterone (dehydroepiandrosterone, DHEA) on sexual dysfunction in postmenopausal women. J Sex Med. 2014 Jul;11(7):1766-85. doi: 10.1111/jsm.12517. Epub 2014 Apr 28. PMID 24774442
- [Result] Portman DJ, Labrie F, Archer DF, Bouchard C, Cusan L, Girard G, Ayotte N, Koltun W, Blouin F, Young D, Wade A, Martel C, Dube R; other participating members of VVA Prasterone Group. Lack of effect of intravaginal dehydroepiandrosterone (DHEA, prasterone) on the endometrium in postmenopausal women. Menopause. 2015 Dec;22(12):1289-95. doi: 10.1097/GME.0000000000000470. PMID 25968836
- [Result] Labrie F. Intravaginal DHEA, by a strictly local action, exerts beneficial effects on both vaginal atrophy symptoms and sexual dysfunction. Horm Mol Biol Clin Investig. 2010 Dec 1;4(1):499-507. doi: 10.1515/HMBCI.2010.064. PMID 25961226
- [Result] Martel C, Labrie F, Archer DF, Ke Y, Gonthier R, Simard JN, Lavoie L, Vaillancourt M, Montesino M, Balser J, Moyneur E; other participating members of the Prasterone Clinical Research Group. Serum steroid concentrations remain within normal postmenopausal values in women receiving daily 6.5mg intravaginal prasterone for 12 weeks. J Steroid Biochem Mol Biol. 2016 May;159:142-53. doi: 10.1016/j.jsbmb.2016.03.016. Epub 2016 Mar 10. PMID 26972555

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 403 subjects were screened at 8 medical/research sites located in the US (2 centers) and Canada (6 centers) and 218 subjects were randomized. The first subject first visit was on 28-JUN-2007 and the last subject last visit was on 23-MAY-2008.
Groups:
- 0.50% DHEA: DHEA (0.50%): Vaginal suppository containing 0.50% (6.5 mg) DHEA; daily dosing with one suppository for 12 weeks.
- 1.00% DHEA: DHEA (1.00%): Vaginal suppository containing 1.0% (13 mg) DHEA; daily dosing with one suppository for 12 weeks.
Period: Overall Study
Arm/Group | Placebo | 0.25% DHEA | 0.50% DHEA | 1.00% DHEA
Started | 54 | 54 | 56 | 54
Safety Population | 54 | 53 | 56 | 54
ITT Population | 53 | 53 | 56 | 54
Completed | 48 | 48 | 52 | 51
Not Completed | 6 | 6 | 4 | 3
Not completed — Adverse Event | 2 | 4 | 2 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 3 | 2 | 0 | 1
Not completed — Left the city/Lost medication | 1 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Baseline Analysis Population corresponds to the Safety Population which includes all subjects who received any amount of prasterone or placebo, and who have any safety information available.
Groups:
- 0.50% DHEA: DHEA (0.50%): Vaginal suppository containing 0.5% (6.5 mg) DHEA; daily dosing with one suppository for 12 weeks.
- 1.00% DHEA: DHEA (1.00%): Vaginal suppository containing 1.00% (13 mg) DHEA; daily dosing with one suppository for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo | 0.25% DHEA | 0.50% DHEA | 1.00% DHEA | Total
Number analyzed (Participants) | 54 | 53 | 56 | 54 | 217
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.00 (5.40) | 57.68 (6.31) | 58.45 (5.55) | 59.44 (4.63) | 58.65 (5.50)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 54 | 53 | 56 | 54 | 217
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White Caucasian | 50 | 51 | 54 | 53 | 208
  Black or African American | 0 | 0 | 0 | 0 | 0
  Asian | 3 | 1 | 1 | 1 | 6
  Other | 1 | 1 | 1 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Co-primary Endpoint: Change From Baseline to Week 12 of Vaginal Cell Maturation (Percentage of Parabasal Cells)
Description: The percentage of parabasal cells was determined from the vaginal smears collected during the study. A 100-cell count was performed by a central laboratory to classify cells as parabasal (P) (including basal), intermediate (I), and superficial (S) squamous cell types. Data obtained at Baseline and Week 12 as well as the change from Baseline to Week 12 are presented.
Time Frame: Baseline and Week 12
Population: The analysis was performed on a subgroup of the ITT Population (defined as all treated subjects with a baseline and at least one post-baseline efficacy assessment) who had self-identified moderate/severe pain at intercourse (Dyspareunia) as their Most Bothersome Symptom of VVA and had ≤ 5% of Superficial Cells and a vaginal pH > 5 on Day 1.
Measure: Mean (Standard Error); unit: percentage of parabasal cells
Arm/Group | Placebo | 0.25% DHEA | 0.50% DHEA | 1.00% DHEA
Number analyzed (Participants) | 26 | 29 | 30 | 29
percentage of parabasal cells
  Baseline | 46.7 (8.64) | 65.5 (6.92) | 53.4 (7.49) | 61.8 (6.88)
  Week 12 | 47.8 (7.52) | 16.9 (3.66) | 11.0 (3.43) | 6.90 (1.77)
  Change from Baseline | 1.1 (3.62) | -48.6 (6.78) | -42.4 (7.36) | -54.9 (6.60)

2. Primary Outcome: Co-primary Endpoint: Change From Baseline to Week 12 of Vaginal Cell Maturation (Percentage of Superficial Cells)
Description: The percentage of superficial cells was determined from the vaginal smears collected during the study. A 100-cell count was performed by a central laboratory to classify cells as parabasal (P) (including basal), intermediate (I), and superficial (S) squamous cell types. Data obtained at Baseline and Week 12 as well as the change from Baseline to Week 12 are presented.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Error); unit: percentage of superficial cells
Arm/Group | Placebo | 0.25% DHEA | 0.50% DHEA | 1.00% DHEA
Number analyzed (Participants) | 26 | 29 | 30 | 29
percentage of superficial cells
  Baseline | 0.6 (0.2) | 0.4 (0.15) | 0.4 (0.11) | 0.4 (0.16)
  Week 12 | 0.5 (0.19) | 5.7 (1.33) | 5.2 (1.19) | 6.5 (1.53)
  Change from Baseline | -0.1 (0.23) | 5.3 (1.39) | 4.8 (1.20) | 6.1 (1.54)

3. Primary Outcome: Co-primary Endpoint: Change From Baseline to Week 12 of Vaginal pH.
Description: A pH strip was applied directly to the lateral wall of the vagina using forceps. The change in color of the pH indicator strip was compared to the color chart for pH evaluation. The corresponding pH value (with one decimal) was recorded. Data obtained at Baseline and Week 12 as well as the change from Baseline to Week 12 are presented.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Error); unit: pH
Arm/Group | Placebo | 0.25% DHEA | 0.50% DHEA | 1.00% DHEA
Number analyzed (Participants) | 26 | 29 | 30 | 29
pH
  Baseline | 6.5 (0.13) | 6.6 (0.10) | 6.6 (0.09) | 6.5 (0.11)
  Week 12 | 6.0 (0.22) | 5.5 (0.19) | 5.2 (0.17) | 5.1 (0.12)
  Change from Baseline | -0.5 (0.16) | -1.1 (0.16) | -1.5 (0.18) | -1.4 (0.15)

4. Primary Outcome: Co-primary Endpoint: Change From Baseline to Week 12 of Self-assessment of the Most Bothersome Symptom Dyspareunia
Description: The severity of dyspareunia was evaluated by a questionnaire. The severity of dyspareunia recorded as none, mild, moderate or severe was analyzed using the score values of 0, 1, 2 or 3, respectively. Data obtained at Baseline and Week 12 as well as the change from Baseline to Week 12 are presented.
Time Frame: Baseline and Week 12
Population: The analysis was performed on a subgroup of the ITT Population (defined as all treated subjects with a baseline and at least one post-baseline efficacy assessment) who had self-identified moderate/severe dyspareunia as their Most Bothersome Symptom of vulvovaginal atrophy (VVA) and had ≤ 5% of Superficial Cells and a vaginal pH > 5 on Day 1.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 0.25% DHEA | 0.50% DHEA | 1.00% DHEA
Number analyzed (Participants) | 26 | 29 | 30 | 29
units on a scale
  Baseline | 2.8 (0.08) | 2.8 (0.08) | 2.7 (0.08) | 2.6 (0.09)
  Week 12 | 2.3 (0.18) | 1.4 (0.22) | 1.1 (0.22) | 1.2 (0.20)
  Change from Baseline | -0.4 (0.16) | -1.3 (0.20) | -1.6 (0.21) | -1.4 (0.18)

5. Secondary Outcome: Change From Baseline to Week 12 of Vaginal Secretions
Description: To evaluate the aspect of the vaginal mucosa and the local tolerance to DHEA suppository, the vaginal secretions (one of the four main signs of vaginal atrophy) evaluated by the physician/gynecologist as corresponding to none, mild, moderate, or severe atrophy were analyzed using the score values of 1, 2, 3 and 4, respectively. Data obtained at Baseline and Week 12 as well as the change from Baseline to Week 12 are presented.
Time Frame: Baseline and Week 12
Population: The analysis was performed on the ITT Population defined as all treated subjects (who received at least one dose) with a baseline and at least one post-baseline efficacy assessment.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 0.25% DHEA | 0.50% DHEA | 1.00% DHEA
Number analyzed (Participants) | 53 | 53 | 56 | 54
units on a scale
  Baseline | 3.1 (0.09) | 3.1 (0.09) | 3.2 (0.09) | 3.0 (0.08)
  Week 12 | 2.7 (0.12) | 1.9 (0.10) | 1.8 (0.12) | 1.5 (0.09)
  Change from Baseline | -0.4 (0.10) | -1.2 (0.12) | -1.4 (0.13) | -1.4 (0.11)

6. Secondary Outcome: Change From Baseline to Week 12 of Vaginal Epithelial Integrity
Description: To evaluate the aspect of the vaginal mucosa and the local tolerance to DHEA suppository, the vaginal epithelial integrity (one of the four main signs of vaginal atrophy) evaluated by the physician/gynecologist as corresponding to none, mild, moderate, or severe atrophy was analyzed using the score values of 1, 2, 3 and 4, respectively. Data obtained at Baseline and Week 12 as well as the change from Baseline to Week 12 are presented.
Time Frame: Baseline and Week 12
Population: as for outcome 5
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 0.25% DHEA | 0.50% DHEA | 1.00% DHEA
Number analyzed (Participants) | 53 | 53 | 56 | 54
units on a scale
  Baseline | 2.8 (0.13) | 2.7 (0.12) | 2.8 (0.11) | 2.7 (0.11)
  Week 12 | 2.4 (0.13) | 1.7 (0.11) | 1.5 (0.10) | 1.4 (0.09)
  Change from Baseline | -0.4 (0.12) | -1.0 (0.14) | -1.3 (0.12) | -1.3 (0.11)

7. Secondary Outcome: Change From Baseline to Week 12 of Vaginal Epithelial Surface Thickness
Description: To evaluate the aspect of the vaginal mucosa and the local tolerance to DHEA suppository, the vaginal epithelial surface thickness(one of the four main signs of vaginal atrophy) evaluated by the physician/gynecologist as corresponding to none, mild, moderate, or severe atrophy was analyzed using the score values of 1, 2, 3 and 4, respectively. Data obtained at Baseline and Week 12 as well as the change from Baseline to Week 12 are presented.
Time Frame: Baseline and Week 12
Population: as for outcome 5
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 0.25% DHEA | 0.50% DHEA | 1.00% DHEA
Number analyzed (Participants) | 53 | 53 | 56 | 54
units on a scale
  Baseline | 3.0 (0.10) | 2.9 (0.08) | 3.1 (0.09) | 3.0 (0.08)
  Week 12 | 2.6 (0.12) | 1.9 (0.11) | 1.8 (0.11) | 1.6 (0.10)
  Change from Baseline | -0.4 (0.10) | -1.0 (0.12) | -1.3 (0.12) | -1.4 (0.12)

8. Secondary Outcome: Change From Baseline to Week 12 of Vaginal Color
Description: To evaluate the aspect of the vaginal mucosa and the local tolerance to DHEA suppository, the vaginal color (one of the four main signs of vaginal atrophy) evaluated by the physician/gynecologist as corresponding to none, mild, moderate, or severe atrophy was analyzed using the score values of 1, 2, 3 and 4, respectively. Data obtained at Baseline and Week 12 as well as the change from Baseline to Week 12 are presented.
Time Frame: Baseline and Week 12
Population: as for outcome 5
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 0.25% DHEA | 0.50% DHEA | 1.00% DHEA
Number analyzed (Participants) | 53 | 53 | 56 | 54
units on a scale
  Baseline | 3.1 (0.09) | 3.0 (0.10) | 3.1 (0.09) | 3.1 (0.07)
  Week 12 | 2.7 (0.11) | 2.0 (0.12) | 1.8 (0.11) | 1.6 (0.10)
  Change from Baseline | -0.5 (0.11) | -1.0 (0.13) | -1.3 (0.14) | -1.5 (0.12)

ADVERSE EVENTS:
Time Frame: From Baseline to Week 12 (+ 30-day follow-up period after last dose)
Arm/Group | Placebo | 0.25% DHEA | 0.50% DHEA | 1.00% DHEA
Serious Adverse Events (participants affected / at risk) | 0/54 | 1/53 | 1/56 | 0/54
Other Adverse Events (participants affected / at risk) | 34/54 | 32/53 | 46/56 | 39/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=54) | 0.25% DHEA (N=53) | 0.50% DHEA (N=56) | 1.00% DHEA (N=54)
Cholecystectomy (Surgical and medical procedures) | 0 | 1 | 0 | 0
Appendicetomy (Surgical and medical procedures) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=54) | 0.25% DHEA (N=53) | 0.50% DHEA (N=56) | 1.00% DHEA (N=54)
Abdominal pain (Gastrointestinal disorders) | 4 | 2 | 3 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 2 | 4 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 7 | 1
Fatigue (General disorders) | 1 | 3 | 4 | 5
Headache (Nervous system disorders) | 3 | 6 | 6 | 4
Hot flush (Reproductive system and breast disorders) | 4 | 2 | 4 | 4
Nasopharyngitis (Infections and infestations) | 5 | 6 | 4 | 4
Vaginal discharge (Reproductive system and breast disorders) | 3 | 4 | 6 | 2
Vulvovaginal burning sensation (Reproductive system and breast disorders) | 4 | 1 | 3 | 4
Vulvovaginal pruritus (Reproductive system and breast disorders) | 3 | 4 | 5 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators shall provide to the SPONSOR 30 days prior to submission all documents for publication, presentation, etc that report any trial results. The SPONSOR shall have editorial rights on documents and the right to review/comment with regard to (1) proprietary information, (2) accuracy of the information, (3) correctness of the scientific evaluation/conclusions and (4) to ensure that the information is fairly balanced and in compliance with regulations.